CLINICAL TRIAL: NCT07230106
Title: A Phase II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics, and Efficacy of HS-20093 or SHR2554 Tablets in Combination With Novel Hormonal Agents in Participants With Metastatic Prostate Cancer
Brief Title: A Study of SHR3680, HS-20093 and SHR2554 in Subjects With Prostate Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR3680-205
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Injections; abiraterone; enzalutamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 Group (Experimental)
  Interventions: Drug: HS-20093 for Injection; Drug: SHR3680 Tablet; Drug: Abiraterone Tablet
- Cohort 2 Group (Experimental)
  Interventions: Drug: SHR3680 Tablet; Drug: SHR2554 Tablet; Drug: Enzalutamide Tablet; Drug: Darotamine Capsule

INTERVENTIONS:
Drug: HS-20093 for Injection — HS-20093 for injection.
  Arms: Cohort 1 Group
Drug: SHR3680 Tablet — SHR3680 tablet.
Drug: Abiraterone Tablet — Abiraterone tablet.
  Arms: Cohort 1 Group
Drug: SHR2554 Tablet — SHR2554 tablet.
  Arms: Cohort 2 Group
Drug: Enzalutamide Tablet — Enzalutamide tablet.
  Arms: Cohort 2 Group
Drug: Darotamine Capsule — Darotamine capsule.
  Arms: Cohort 2 Group

SUMMARY:
This is a phase II, multicentre clinical study investigating HS-20093 or SHR2554 in combination with a Novel Hormonal Agent (NHA) for advanced prostate cancer. The trial comprises two cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this clinical study, understand the research procedures, and are able to provide written informed consent.
2. Aged 18 to 80 years (inclusive), male.
3. ECOG performance status of 0 or 1.
4. Expected survival time ≥12 weeks.
5. Histologically or cytologically confirmed prostate adenocarcinoma, with no features of neuroendocrine carcinoma or small cell carcinoma.
6. Able to provide sufficient tumor tissue samples for retrospective genetic testing.
7. Ongoing Androgen Deprivation Therapy (ADT) throughout the study period, i.e., continuous treatment with a GnRH agonist or antagonist (chemical castration) or prior bilateral orchiectomy (surgical castration).
8. PSA level ≥1 ng/ml at screening.
9. Adequate organ function levels at baseline assessment.
10. Male participants with female partners of childbearing potential must agree to refrain from sperm donation and use effective contraception from the time of signing the informed consent form until 4.5 months after the last dose of HS-20093 or 3 months after the last dose of other study treatments, whichever is later.

Exclusion Criteria:

1. Known hypersensitivity or intolerance to the investigational drug(s) or their excipients.
2. Adverse events from prior anti-tumor therapy have not recovered to Grade ≤1 as per CTCAE v5.0.
3. Administration of estrogen, progesterone, or 5-alpha reductase inhibitors within 28 days prior to enrollment.
4. Administration of herbal medicines known to have anti-prostate cancer or PSA-lowering effects within 14 days prior to enrollment.
5. Major surgery within 28 days prior to enrollment; palliative radiotherapy within 14 days prior to enrollment; or traumatic minor surgery within 7 days prior to enrollment.
6. Pathological fractures in critical locations, spinal cord compression, etc., within the recent 6 months.
7. Non-healing wounds, untreated fractures, or severe bone damage due to metastatic disease.
8. Poorly controlled tumor-related pain.
9. Dysphagia or other conditions significantly affecting drug absorption.
10. Known central nervous system metastases or primary brain tumors.
11. Significant pericardial, pleural, or peritoneal effusion requiring intervention.
12. Severe cardiovascular or cerebrovascular diseases.
13. Moderate to severe pulmonary disease significantly affecting respiratory function.
14. Poorly controlled diabetes.
15. Serious active infections within 14 days prior to enrollment.
16. Active Hepatitis B, Hepatitis C, HIV, or immunodeficiency diseases.
17. History of other malignancies within 5 years prior to enrollment.
18. Any other condition deemed by the investigator to potentially affect the study.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: 6-month undetectable Prostate Specific Antigen (PSA) rate. | 6 months.
Cohort 2: Prostate Specific Antigen (PSA) response rate. | About 2 years.
Cohort 2: Adverse events (AEs). | About 2 years.
Cohort 2: Dose-limiting toxicity (DLT). | About 28 days.

SECONDARY OUTCOMES:
Radiographic Progression-Free Survival (rPFS). | About 2 years.
Time to Prostate Specific Antigen (PSA) progression. | About 2 years.
Time to Next Symptomatic Skeletal Event (SSE). | About 2 years.
Time to Next Antineoplastic Therapy (TTNT). | About 2 years.
Objective response rate (ORR). | About 2 years.
Cohort 1: Adverse events (AEs). | About 2 years.
Disease control rate (DCR). | About 2 years.
Duration of response (DoR). | About 2 years.
Overall Survival (OS). | About 2 years.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided